CLINICAL TRIAL: NCT04379882
Title: Feasibility Study Evaluating the Silva Module During the Anaesthesiology Consultation Before an Elective Surgery
Acronym: Silva
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Decision of alternative research to be performed
Sponsor: Oncomfort (Industry)
Collaborators: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OC32 Silva
Record Dates: First submitted 2020-04-17; First posted 2020-05-08 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Preoperative Anxiety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital sedation (Experimental): 30 minutes Silva module
  Interventions: Device: Digital Sedation (Silva)

INTERVENTIONS:
Device: Digital Sedation (Silva) — Use of Digital Sedation (virtual reality associated with psychological interventions) for preoperative anxiety management

SUMMARY:
In this feasibility study, feasibility, acceptability and an initial clinical efficacy of the new module of Hypnosis and Virtual Reality (or Digital Sedation), Silva, will be evaluated. This feasibility study meets objectives of Oncomfort's design validation and design verification steps. Silva will be tested on a sample of 10 patients in the environment where the product is intended to be used, a hospital environment. If results do not fit with user needs, design will be adapted according to results and a new phase of design validation will be implemented. The Silva module is a Digital Sedation module designed for management of pain and anxiety in perioperative patients.

DETAILED DESCRIPTION:
Subjects will be recruited during the anaesthesiology consultation preparing to an elective surgery.

First, subject will be asked to self-assess anxiety and comfort. In order to evaluate anxiety, subject will use a 0-10 rating Visual Analogue Scale (VAS) where 0 = no anxiety at all, and 10= the worst imaginable anxiety. The same scale will be used to measure the level of comfort where 0 means no comfort at all and 10 very comfortable.

Subject should be positioned laying on a reclining chair during the session. This session will last for 30 minutes. After the experiment, participants will be asked to rate anxiety, level of comfort, level of immersion and dissociation.

Several questions will be asked to the patient to evaluate his/ her experience, the Silva module, and the sensations experienced.

The study will be ended by an evaluation of adverse event (AE) and the evaluation of the caregivers.

ELIGIBILITY:
Inclusion Criteria:

• Subject more than 18 years old

Exclusion Criteria:

* Deaf subject
* Blind
* Non-proficiency in French (Module language)
* Psychiatric disorder
* Head or face wounds
* Neurological disease
* Chronic pain and/or chronic analgesics consumption
* Medication affecting the autonomic nervous system
* Dizziness

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-10 (Estimated); Primary Completion 2020-12-10 (Estimated); Study Completion 2020-12-20 (Estimated)

PRIMARY OUTCOMES:
Evaluate the acceptability and the patient's qualitative reported experience of Silva | Day 1 of the intervention
  questionnaire

SECONDARY OUTCOMES:
Evaluate Anxiety | Day 1 of the intervention
  questionnaire VAS 0 (no anxiety)- 10 (max anxiety)
Evaluate Comfort | Day 1 of the intervention
  questionnaire VAS 0 (extreme discomfort)- 10 (extreme comfort)
Evaluation of agreeability of the Digital Sedation session | Day 1 of the intervention
  questionnaire VAS (0-10) 0: not agreeable, 10: extremely agreeable

IPD SHARING:
Plan to Share IPD: No